CLINICAL TRIAL: NCT00443352
Title: A Single-Center, Open Label Pilot Study Examining The Use Of Duloxetine In The Prevention Of Episodic Migraine
Brief Title: A Research Study Examining The Use Of Duloxetine In The Prevention Of Migraine Headache
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Protocol #: F1J-MC-I
Record Dates: First submitted 2007-03-05; First posted 2007-03-06 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-04

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Duloxetine (Experimental): Duloxetine 120mg daily for 12 weeks.
  Interventions: Drug: duloxetine

INTERVENTIONS:
Drug: duloxetine — Duloxetine: 120 mg. daily or maximum tolerated dose (minimum: 60 mg per day)
  Other Names: Cymbalta

SUMMARY:
This is a single-center, open-label, pilot trial to collect and evaluate data on the safety and efficacy of duloxetine in the preventive treatment of subjects experiencing episodic migraine headaches. Following a 28-day baseline period, qualifying subjects will be entered into an 84-day treatment period. Subjects will be titrated over the first four weeks to a dose of 120mg or their maximally tolerated dose (MTD). The dose adjustments will be based on individual subject response and/or subject's tolerability. Subjects will maintain a daily diary capturing detailed information on migraine headache days.

DETAILED DESCRIPTION:
Pharmacologic therapy of migraine headaches can be divided into two types: acute treatment and prophylactic treatment. Acute headache medication is intended to relieve the pain and disability of an acute attack and stop its progression. Prophylactic (preventive) headache therapy is generally given daily, even in the absence of headache, to reduce the frequency and perhaps the severity of anticipated attacks. Subjects who experience recurring migraine attacks which significantly interfere with the subject's daily routine despite acute treatment, may warrant chronic prophylactic treatment.

Duloxetine may be an important treatment option for millions of unsuccessfully treated migraine patients and therefore warrants further study. Considering this, we propose a single-center, open-label pilot trial to collect and evaluate data on the safety and efficacy of duloxetine in the preventive treatment of subjects with episodic migraine headaches. The results of this pilot trial will provide preliminary insight into the clinical role duloxetine may play in the treatment of headache, as well as provide a basis for future well-controlled trials of this medication.

This is a single-center, open-label, pilot trial to collect and evaluate data on the safety and efficacy of duloxetine in the preventive treatment of subjects experiencing episodic migraine headaches. Following a 28-day baseline period, qualifying subjects will be entered into an 84-day treatment period. Subjects will be titrated over the first four weeks to a dose of 120mg or their maximally tolerated dose (MTD). The dose adjustments will be based on individual subject response and/or subject's tolerability. Subjects will maintain a daily diary capturing detailed information on migraine headache days.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female between the ages of 18 and 65, inclusive
* Subject has an IHS diagnosis of migraine with or without aura for at least one-year prior to screening
* Subject has experienced between 4 and 10 migraine headaches per month (inclusive) over the past six months, with at least 24 hours separating attacks
* Subject has less than 15 total headache days per month
* Subject is able to differentiate migraine attacks from other headache types, if applicable
* Subjects daily medications (for any indication) have remained at a stable dose for the 60 days preceding screening
* Subject is using or agrees to use for the duration of participation a medically acceptable form of contraception (as determined by investigator and mutually agreed upon with patient), if female of child-bearing potential
* Subjects currently taking a single agent for the prevention of migraine must be on a stable dose (unchanged for 2 months) prior to study entry
* Subject has negative urine pregnancy test prior to study entry, if female of child-bearing potential
* Subject is able to understand and comply with all study requirements
* Subject provides written informed consent prior to any screening procedures being conducted

EXCLUSION CRITERIA:

* Subjects with onset of migraine after 50 years of age
* Subjects who have been previously treated or are currently being treated with duloxetine
* Subjects who have failed greater than 3 adequate trials of other medications the prevention of migraine, as determined by investigator
* Subjects who have a known hypersensitivity to duloxetine or any of the inactive ingredients
* Subject has taken any medication which has been shown to be effective for migraine prophylaxis, on a daily basis within the 4 weeks prior to screening or at any time during participation in the study, for any indication.
* Subjects with a history of significant drug or alcohol abuse within the past year
* Subjects with major depressive disorder or who have had a suicidal ideation in the 3 months prior to screening or have a history of attempted suicide
* Subjects who have a Beck Depression Inventory score of > 18 at screening
* Subjects who have > 0 on question number 9 of Beck Depression Inventory (Suicidal Thoughts or Wishes question)
* Subjects who have participated in an investigational drug trial in the 30 days prior to the screening visit
* Subjects with a current or history of a hepatic or renal disorder
* Subjects with uncontrolled narrow angle glaucoma
* Subjects who have experienced significant side effects from two different SSRI and/or SNRI therapies, as determined by investigator
* Subjects with uncontrolled restless legs syndrome, as determined by investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William B. Young, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Jefferson Headache Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Duloxetine
Started | 27
Completed | 22
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- Duloxetine Completers: duloxetine: Duloxetine: 120 mg. daily or maximum tolerated dose (minimum: 60 mg per day)
Arm/Group | Duloxetine Completers
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Frequency of Migraine Days During the Last 28 Day Interval of the Treatment Period as Compared to the 28 Day Baseline Period.
Description: Change in frequency of migraine days from day -28 to day 0 (28 days) was compared to frequency of migraine days from day 56-84 (final 28 days of study).
Time Frame: Change in frequency of migraine days from day -28 to day 0 (28 days) was compared to frequency of migraine days from day 56-84 (final 28 days of study).
Population: Number of participants for analysis was modified intention to treat - anyone who took at least one dose of duloxetine
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Duloxetine
Number analyzed (Participants) | 27
days | 4.5 (3.4)

ADVERSE EVENTS:
Arm/Group | Duloxetine
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 15/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=27)
Dry mouth (General disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 8 (8)
Fatigue (General disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
This trial was uncontrolled. Five of the 27 subjects did not complete.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes